CLINICAL TRIAL: NCT01495260
Title: A Clinical Trial for Adrenomyeloneuropathy (AMN): Validation of Biomarkers of Oxidative Stress, and Efficacy, Tolerance and Safety of a Mixture of the Antioxidants N-acetylcysteine, Lipoic Acid and Vitamin E
Brief Title: A Clinical Trial for AMN: Validation of Biomarkers of Oxidative Stress, Efficacy and Safety of a Mixture of Antioxidants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pujol, Aurora, M.D. (Individual)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government); Fundacion Hesperia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XAMNANTIOXAP2010
Record Dates: First submitted 2011-11-28; First posted 2011-12-19 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2016-09

CONDITIONS: Adrenomyeloneuropathy
Keywords: XALD; AMN
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Acetylcysteine; Thioctic Acid; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N-acetylcysteine, lipoic acid and vitamin E (Experimental): Two Dose titration design
  Interventions: Drug: N-acetylcysteine; Drug: lipoic acid; Drug: vitamin E

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine, 800-2400 mg daily for 2 months
Drug: lipoic acid — lipoic acid, 300-600 mg daily for 2 months
Drug: vitamin E — vitamin E, 150-300 mg daily for 2 months

SUMMARY:
X-linked adrenoleukodystrophy is a rare, demyelinating and neurodegenerative disorder, due to a loss of function of a fatty acid transporter, the peroxisomal ABCD1protein. Its more frequent phenotype, the adrenomyeloneuropathy in adults, is characterized by axonal degeneration in spinal cord, spastic paraparesis and a disabling peripheral neuropathy. Actually, there is no efficient treatment for the disease. Our work in the last twelve years dissecting the physiopathological basis of the disorder has uncovered an involvement of the oxidative stress early in the neurodegenerative cascade. In a preclinical trial we have identified an antioxidant cocktail that efficiently reverse the clinical symptoms and the axonal degeneration in the mouse model for the disease. We propose the translation of the results to an open trial to test the tolerance and effectiveness of these drugs in the correction of the previously identified oxidative lesion biomarkers, as a first step to a randomized versus placebo, multicentric and international trial. You will be clinically explored and assessed in the Hospital Universitari of Bellvitge (HUB) using clinical scales for spasticity, disability, electroneurogram and cranial and spinal Nuclear Magnetic resonance (NMR). The information will be collected in a data base that will be of great value to improve the present attention and the future follow-up to facilitate your inclusion in therapeutic randomized, double blind, against placebo clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic AMN patients,
* 18-64 years old,
* male and female,
* clinically and biochemically diagnosed;
* females must be obligated heterozygotes or must have gene mutation identified.

Exclusion Criteria:

* Pregnant and lactation in females,
* Cerebral inflammatory disease with cognitive disorder, and/or
* need the help of two walking sticks,
* epilepsy,
* hypersensibility to cysteine related compounds,
* transaminases 2 fold up normal values.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
oxidative lesion biomarkers | 12 months
  oxidative lesion biomarkers: protein, DNA and peroxidation biomarkers

SECONDARY OUTCOMES:
clinical parameters | 2, 6 and 12 months
  spasticity, disability,electroneurograms and evocated potentials. Cranial and spinal NMR will be done at the beginning and the end of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Lopez-Erauskin J, Fourcade S, Galino J, Ruiz M, Schluter A, Naudi A, Jove M, Portero-Otin M, Pamplona R, Ferrer I, Pujol A. Antioxidants halt axonal degeneration in a mouse model of X-adrenoleukodystrophy. Ann Neurol. 2011 Jul;70(1):84-92. doi: 10.1002/ana.22363. PMID 21786300
- [Background] Galino J, Ruiz M, Fourcade S, Schluter A, Lopez-Erauskin J, Guilera C, Jove M, Naudi A, Garcia-Arumi E, Andreu AL, Starkov AA, Pamplona R, Ferrer I, Portero-Otin M, Pujol A. Oxidative damage compromises energy metabolism in the axonal degeneration mouse model of X-adrenoleukodystrophy. Antioxid Redox Signal. 2011 Oct 15;15(8):2095-107. doi: 10.1089/ars.2010.3877. Epub 2011 Jun 8. PMID 21453200
- [Derived] Parameswaran J, Goicoechea L, Planas-Serra L, Pastor A, Ruiz M, Calingasan NY, Guilera C, Aso E, Boada J, Pamplona R, Portero-Otin M, de la Torre R, Ferrer I, Casasnovas C, Pujol A, Fourcade S. Activating cannabinoid receptor 2 preserves axonal health through GSK-3beta/NRF2 axis in adrenoleukodystrophy. Acta Neuropathol. 2022 Aug;144(2):241-258. doi: 10.1007/s00401-022-02451-2. Epub 2022 Jul 1. PMID 35778568
- [Derived] Casasnovas C, Ruiz M, Schluter A, Naudi A, Fourcade S, Veciana M, Castaner S, Alberti A, Bargallo N, Johnson M, Raymond GV, Fatemi A, Moser AB, Villarroya F, Portero-Otin M, Artuch R, Pamplona R, Pujol A. Biomarker Identification, Safety, and Efficacy of High-Dose Antioxidants for Adrenomyeloneuropathy: a Phase II Pilot Study. Neurotherapeutics. 2019 Oct;16(4):1167-1182. doi: 10.1007/s13311-019-00735-2. PMID 31077039
- See also: The Neurometabolic Diseases Lab, led by ICREA Research Professor Aurora Pujol, is integrated in the Neurosciences Area of IDIBELL. — http://www.neurometabolic-lab.org/
- See also: Related Info — http://www.idibell.cat/
- See also: Related Info — http://www.bellvitgehospital.cat/